CLINICAL TRIAL: NCT00869583
Title: Enlace: A Partnership to Promote Physical Activity Among Mexican Immigrant Women
Brief Title: Increasing Physical Activity Among Mexican American Women (The Enlace Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 642; R21HL087765 (NIH); 7R21HL087765 (NIH)
Record Dates: First submitted 2009-03-25; First posted 2009-03-26 (Estimated); Last update posted 2019-08-16 (Actual); Status verified 2014-01

CONDITIONS: Obesity; Heart Diseases
Keywords: Women; Physical Activity; Hispanic; Overweight
MeSH Terms: conditions — Obesity; Heart Diseases; Motor Activity; Overweight

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Participants will immediately take part in the physical activity program.
  Interventions: Behavioral: Physical Activity Program
- 2 (No Intervention)

INTERVENTIONS:
Behavioral: Physical Activity Program — Participants will receive counseling from a community health educator that will focus on the importance of increasing physical activity. Participants will be encouraged to engage in moderate physical activity (3.0 to 6.0 metabolic equivalents [METS]) for 30 minutes on 5 or more days per week. Participants will be encouraged to start their physical activity program slowly and to gradually increase both frequency and intensity to meet the study goal (e.g., beginning with three sessions per week for 15 minutes and building up to five sessions per week for 30 minutes by Week 12). They will receive educational materials and telephone calls or visits from health educators on a monthly basis for 6 months.
  Arms: 1

SUMMARY:
Obesity is a serious health problem among Mexican American women. Obesity combined with a lack of physical activity can increase the risk for several diseases, including heart disease. This study will evaluate a program that aims to increase physical activity levels among women of Mexican origin in Columbia, South Carolina and the Lower Rio Grande Valley of Texas.

DETAILED DESCRIPTION:
Mexican American women in the United States are more likely to live a sedentary lifestyle than women of other ethnic groups. As a result, obesity affects Mexican American women at a high rate. Obesity and a lack of physical activity are risk factors for many diseases, including heart disease, diabetes, and certain types of cancers. Increasing physical activity can lead to weight loss and lower the risk of developing these diseases. This study represents a partnership between the University of South Carolina, the South Carolina Hispanic Latino Health Coalition, and the University of Texas Health Sciences Center at San Antonio (UTHSCSA) Regional Academic Health Center in the Lower Rio Grande Valley of Texas. Study researchers from these institutions will first conduct interviews and focus groups and then develop a program aimed at encouraging moderately intense physical activity among Mexican American women. Next, the study will evaluate the effectiveness of that program at increasing physical activity levels and promoting weight loss among Mexican American women in Columbia, South Carolina and the Lower Rio Grande Valley of Texas.

This study will enroll Mexican American women. Participants will be randomly assigned to either immediately take part in the physical activity program or take part in the program at the end of the 6-month study. At baseline, all participants will receive home visits from study staff. During these visits, participants will undergo weight, height, and waist measurements. Participants will also complete questionnaires to assess their medical history and physical activity habits. For 1 week after the study visit, participants will wear a physical activity monitor and keep an activity diary. Participants who are assigned to immediately take part in the physical activity program will receive counseling from a community health educator that will focus on the importance of changing physical activity habits. They will be encouraged to partake in 30 minutes of daily physical activity for at least 5 days a week. Each month, participants will receive educational materials and telephone calls or visits from the health educator. Participants will receive a pedometer and will be asked to keep a daily log of their physical activity. At Month 6, all participants will receive another home study visit for repeat baseline testing. At this time, participants who did not take part initially in the physical activity program will start the program. However, they will have no further study visits or evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Self-identifies as being of Mexican origin
* Has a personal telephone
* Resides in the study area and intends to stay in the area for the entire study period
* Able to understand Spanish
* Does not currently meet physical activity level recommendations
* Interested in receiving information on physical activity
* Willing to be assigned to either study group
* Willing to attend the program sessions and complete standardized measurements

Exclusion Criteria:

* Not physically able to participate in a moderate intensity walking program and not able to understand and verbally respond to questions
* Pregnant
* Diabetes
* Uncontrolled hypertension
* Undergoing therapy for life-threatening illnesses (e.g., chemotherapy or radiation therapy)
* Positive (risk) responses on the Physical Activity Readiness Questionnaire (PAR-Q) and subsequent physician disapproval on the Physical Activity Readiness Medical Examination (PAR-Med-X)
* Already gets 5 or more days per week of 30 minutes of moderately intense activity, based on the responses to the six questions concerning frequency and duration of moderately and vigorously intense physical activity from the Behavioral Risk Factor Surveillance Survey

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2009-08; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Moderate to vigorous physical activity (measured by accelerometry and self-report) | Measured at baseline and Month 6

SECONDARY OUTCOMES:
Body mass index | Measured at baseline and Month 6

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Parra-Medina, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (2):
- United States (2):
  - University of South Carolina, Columbia, South Carolina
  - University of Texas Health Science Center San Antonio, San Antonio, Texas

REFERENCES:
- [Background] Parra-Medina D, Hilfinger Messias DK. Promotion of Physical Activity Among Mexican-Origin Women in Texas and South Carolina: An Examination of Social, Cultural, Economic, and Environmental Factors. Quest. 2011 Feb;63(1):100-117. doi: 10.1080/00336297.2011.10483668. PMID 21731409